CLINICAL TRIAL: NCT02292147
Title: Functional Outcome After Cardiac Arrest; Prediction and Prognosis Factors for Patients Awake Within the First 15 Days
Brief Title: Functional Outcome After Cardiac Arrest
Acronym: HANOX
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P111012
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2017-11

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: Cerebral anoxia; Functional outcome
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Descriptive and prognosis study of the functional outcome after cardiac arrest for the patients awake within the first 15 days.

DETAILED DESCRIPTION:
Functional outcome after cerebral anoxia due to cardiac arrest is poorly documented.. Survival after out of hospital cardiac arrest has improved and long term follow up of the patients is not routinely effective. Patients showing sign of awakening very early are considered in a good outcome group. Nevertheless they can experience some restriction and difficulties when they try to return to their premorbid level of functioning.

We aim to study their long term functional outcome and their level of anxiety, depression, quality of life and caregiver burden as well as their general cognitive functioning. Prognosis factors will be studied in the acute phase.

ELIGIBILITY:
Inclusion criteria :

* age 18 to 85
* Out of hospital cardiac arrest ; cardiac arrest in the ER is eligible
* Glasgow Coma Score ≥ 12 within 15 days after onset
* Living in the parisian area

Exclusion criteria :

* no social security
* Neurological condition (multiple sclerosis, parkinson disease, AMS, stroke) priori to the cardiac arrest
* Psychiatric condition (schizophrenia, severe bipolar syndrome, long term neuroleptic medication, autistic spectrum disorders
* Deafness and blindness
* Neoplasia
* Premorbid limitation of autonomy.
* Difficulties in speaking and writing the French language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting an Out of hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Glasgow outcome Scale Extended score | 18 months
  Functional outcome at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Peskine, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Charles-Edouard Luyt, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié salpetriere Hospital, Paris, France

REFERENCES:
- [Result] Peskine A, Cariou A, Hajage D, Deye N, Guerot E, Dres M, Sonneville R, Lafourcade A, Navarro V, Robert H, Azouvi P, Sharshar T, Bayen E, Luyt CE; Hanox Study Group. Long-Term Disabilities of Survivors of Out-of-Hospital Cardiac Arrest: The Hanox Study. Chest. 2021 Feb;159(2):699-711. doi: 10.1016/j.chest.2020.07.022. Epub 2020 Jul 20. PMID 32702410